CLINICAL TRIAL: NCT00673842
Title: Risk Estimation Following Infarction Noninvasive Evaluation - ICD Efficacy
Brief Title: Efficacy of Implantable Defibrillator Therapy After a Myocardial Infarction
Acronym: REFINE-ICD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Calgary (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Alberta Innovation and Science (Other); Medtronic (Industry); GE Healthcare (Industry); Cardiac Arrhythmia Network of Canada (Other); Accelerating Clinical Trials Consortium (Other)
Responsible Party: Principal Investigator, Dr. Derek Exner, Professor and Canada Research Chair in Cardiovascular Clinical Trials, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 21721
Record Dates: First submitted 2008-04-29; First posted 2008-05-07 (Estimated); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Myocardial Infarction; Sudden Death
Keywords: Noninvasive assessment; Holter
MeSH Terms: conditions — Myocardial Infarction; Death, Sudden | interventions — Defibrillators, Implantable

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ICD + Usual Care (Experimental): Implantable Cardioverter Defibrillator + Usual Care
  Interventions: Device: Implantable Cardioverter Defibrillator + Usual Care
- Usual Care (Active Comparator): Usual post-MI care
  Interventions: Other: Usual care

INTERVENTIONS:
Device: Implantable Cardioverter Defibrillator + Usual Care — Any Medtronic approved single chamber or dual chamber implantable cardioverter defibrillator (ICD)
  Other Names: Implantable Cardioverter Defibrillator; ICD
  Arms: ICD + Usual Care
Other: Usual care — Usual post-MI care
  Other Names: Standard medical therapy alone
  Arms: Usual Care

SUMMARY:
This study will assess whether an implantable defibrillator will increase the likelihood of survival in patients who have had a heart attack, have abnormal test results from a 24 hour heart monitor, and who have low normal heart function.

DETAILED DESCRIPTION:
The REFINE ICD trial will assess whether prophylactic ICD therapy, guided by non-invasive risk assessment tools, reduces mortality in MI survivors with better-preserved LV function.

ELIGIBILITY:
Site investigators are responsible for screening. Subjects must meet all inclusion criteria. Subjects with any exclusion criteria will be excluded.

Initial inclusion criteria (eligibility for Holter screening).

* 18 - 80 years old at time of consent
* History of MI ≥ 2 months prior to screening based on ESC/ACCF/AHA/WHF criteria (both STEMI and NSTEMI subjects are eligible)
* Appropriate post-MI management including revascularization where indicated
* No contra-indication for transvenous ICD placement (e.g., mechanical tricuspid valve, known vascular access problems, active sepsis, etc.)
* LVEF 36% - 50% measured at least 40 days after a confirmed MI ≥ 3 months after coronary angioplasty or coronary bypass surgery and within the following time windows:

  * LVEF ≤ 7 months of screening visit if index MI was ≤ 1 year of enrolment
  * LVEF ≤ 13 months of screening visit if index MI was > 1 & < 3 years of enrolment
  * LVEF ≤ 25 months of screening visit if index MI was ≥ 3 years of enrolment
* Proven, necessary or appropriate medications (e.g. beta-blocker, ACE inhibitor / ARB, statin, and anti-platelet)
* In normal sinus rhythm (ECG documented) ≤ 8 weeks prior to the screening Holter
* Written informed consent
* Able and willing to complete the screening Holter, including the six-minute hall walk

Additional inclusion criterion (eligibility for randomization).

* Abnormal HRT & TWA (core lab interpretation) on Holter performed at least 2 months after the index MI and the specified time after coronary revascularization
* In normal sinus rhythm (ECG documented) within 8 weeks prior to the screening Holter
* In normal sinus rhythm for ≥ 18 hours of the 24 hr screening Holter as determined by the study Holter Core Lab

Exclusion criteria (randomization or registry).

* Use of antiarrhythmic drugs
* Clinical indication for permanent pacemaker or a cardiac resynchronization device
* Clinical indication for an ICD or cardiac resynchronization ICD
* Prior implantation of a pacemaker, ICD, or Cardiac Resynchronization device
* Any condition, in the investigator's judgment, that would limit life expectancy to < 12 months
* Chronic renal failure (hemodialysis or peritoneal dialysis)
* Active ischemia that is amenable to revascularization if not previously revascularized
* Participation in another trial that may interfere with the REFINE ICD results.
* Pregnancy
* Inability to comply with the follow-up schedule

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 700 (Estimated)
Dates: Start 2011-04-18 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2024-10-31 (Actual)

PRIMARY OUTCOMES:
Mortality | Minimum of 18 months of follow-up (average follow-up of 5 years).

SECONDARY OUTCOMES:
Cardiac death | Average follow-up 5 years.
Arrhythmic death | Average follow-up 5 years.
Arrhythmic syncope | Average follow-up 5 years.
Appropriate ICD therapies | Average follow-up 5 years.
Quality of life | Average follow-up 5 years.
Inappropriate ICD therapies | Five years (average)

CONTACTS AND LOCATIONS:
Overall Officials: Derek V Exner, MD, MPH, Principal Investigator — University of Calgary
Locations (78):
- United States (29):
  - Heart Center Research LLC, Huntsville, Alabama
  - Colorado Heart and Vascular, Lakewood, Colorado
  - James A Haley Veterans' Center, Tampa, Florida
  - The Heart Group/Deaconess, Evansville, Indiana
  - Iowa Heart Center, West Des Moines, Iowa
  - Delmarva Heart Foundation, Salisbury, Maryland
  - Beth Israel Deaconess, Boston, Massachusetts
  - Washington University Medical School, Saint Louis, Michigan
  - St. John Providence Hospital, Southfield, Michigan
  - Lester E Cox Medical Center, Springfield, Missouri
  - The Valley Hospital, Ridgewood, New Jersey
  - Associated Cardiovascular Consultants/Lourdes Cardiology Services, Voorhees Township, New Jersey
  - North Shore LIJ, New York, New York
  - New York Presbyterian Hospital, New York, New York
  - Northeast Ohio Cardiovascular Specialists, Akron, Ohio
  - The Lindner Research Center, Cincinnati, Ohio
  - Bethesda North Hospital, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - The Ohio State University, Columbus, Ohio
  - Doylestown Cardiology, Doylestown, Pennsylvania
  - University of Pittsburgh Medical Center UPMC Presbyterian, Pittsburgh, Pennsylvania
  - Geisinger Wyoming Valley Medical Center, Wilkes-Barre, Pennsylvania
  - Greenville Hospital System, Greenville, South Carolina
  - St. Thomas Research Institute, Nashville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Amarillo Heart Group, Amarillo, Texas
  - University of Virginia, Charlottesville, Virginia
  - Centra Medical Group, Lynchburg, Virginia
  - Heart Clinics Northwest, Spokane, Washington
- UZ Leuven - Campus Gasthuisberg, Leuven, Belgium
- Canada (27):
  - Libin Cardiovascular Institute of Alberta, Calgary, Alberta
  - Royal Alexandra Hospital, Edmonton, Alberta
  - University of Alberta Hospital, Edmonton, Alberta
  - Fraser Clinical Trials, New Westminster, British Columbia
  - Vancouver General Hospital, Vancouver, British Columbia
  - St. Paul's Hospital/Providence Health Care, Vancouver, British Columbia
  - Victoria Cardiac Arrhythmia Trials, Victoria, British Columbia
  - St. Boniface Hospital, Winnipeg, Manitoba
  - Cardio 1, Winnipeg, Manitoba
  - New Brunswick Heart Centre, Saint John, New Brunswick
  - Queen Elizabeth II Health Sciences Center, Halifax, Nova Scotia
  - Cambridge Cardiac Care Centre, Cambridge, Ontario
  - Hamilton Health Sciences Centre, Hamilton, Ontario
  - University of Western Ontario, London, Ontario
  - Southlake, Newmarket, Ontario
  - Ottawa Heart Institute, Ottawa, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - Toronto General Hospital, Toronto, Ontario
  - Montreal Heart Institute, Montreal, Quebec
  - CHUM, Montreal, Quebec
  - McGill University Health Centre, Montreal, Quebec
  - Centre Hospitalier Universitaire de Sherbrooke (CHUS), Sherbrooke, Quebec
  - Centre Hospitalier Universitaire Regional de Trois-Rivieres (CHRTR), Trois-Rivières, Quebec
  - Prairie Vascular Research Network, Regina, Saskatchewan
  - Royal University Hospital, Saskatoon, Saskatchewan
  - Quebec Heart Institute, Laval
- Finland (2):
  - HUCH Helsinki University Central Hospital, Helsinki
  - University of Oulu, Oulu
- France (3):
  - CHRU Brest - Hôpital de la Cavale Blanche, Brest
  - Hôpital Guillaume et René Laënnec - CHU de Nantes, Nantes
  - Clinique Pasteur, Toulouse
- Universitätsmedizin Göttingen Georg-August-Universität, Göttingen, Germany
- Zala Megyei Kórház, Zalaegerszeg, Hungary
- Italy (3):
  - Azienda Ospedaliera Papa Giovanni XXIII, Bergamo
  - Policlinico Sant' Orsola - Malpighi, Bologna
  - Fondazione IRCCS Policlinico San Matteo, Pavia
- Oslo Universitetssykehus Rikshospitalet, Oslo, Norway
- King Saud University, Riyadh, Saudi Arabia
- Slovak Medical University in Bratislava, Bratislava, Slovakia
- Unitas Hospital, Centurion, South Africa
- Spain (4):
  - Hospital General Universitario de Alicante (HGUA), Alicante
  - Hospital Universitario Clinic de Barcelona, Barcelona
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
- Universitetssjukhuset Örebro, Örebro, Sweden
- United Kingdom (2):
  - Liverpool Heart and Chest Hospital, Liverpool
  - Great Western Hospital NHS Trust, Swindon

IPD SHARING:
Plan to Share IPD: Undecided
uncertain

REFERENCES:
- [Derived] Perkiomaki J, Exner DV, Piira OP, Kavanagh K, Lepojarvi S, Talajic M, Karvonen J, Philippon F, Junttila J, Coutu B, Huikuri H. Heart Rate Turbulence and T-Wave Alternans in Patients with Coronary Artery Disease: The Influence of Diabetes. Ann Noninvasive Electrocardiol. 2015 Sep;20(5):481-7. doi: 10.1111/anec.12244. Epub 2015 Jan 15. PMID 25589197